CLINICAL TRIAL: NCT06826586
Title: Identification of Microplastics in Liver, Stomach, Blood, and Feces of Obese Patients and Their Association Analysis with Macrogenomics and Metabolomics.
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2025-099-01
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Obesity and Overweight
Keywords: microplastics; obesity; macro-genomic; metabolomics
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- obesity group: BMI≧30
  Interventions: Diagnostic Test: Measuring the microplastics

INTERVENTIONS:
Diagnostic Test: Measuring the microplastics — Measuring the type, nature, and abundance of microplastics in stomach, liver, feces, and blood

SUMMARY:
The aim of this study was to identify and quantify microplastics in the stomach, liver, feces, and blood of obese patients to be treated with bariatric surgery by using a variety of advanced analytical techniques to explore the association between obesity and visceral microplastics, and to investigate the effects of microplastics on the visceral microbiota and metabolic profiles of obese patients by combining the macro-genomic and metabolomics approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* BMI ≧30;
* proposed to undergo bariatric surgery and need to remove part of the liver tissue for fatty liver test;
* complete clinical data and basic information;
* willing to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Receive chemotherapy, radiotherapy, immunotherapy;
* have other history of digestive diseases;
* combined with malignant tumors;
* have serious cardiorespiratory insufficiency and other systemic diseases that affect the choice of treatment plan;
* not willing to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with obesity
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in microbial communities | From the diagnosis of obesity, through study completion, an average of 1 year.
  Differences in different microbial communities in the stomach, liver, feces, and blood of obese patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data was not allowed sharing in our ethics committee.